CLINICAL TRIAL: NCT04576091
Title: Phase I Trial of BAY 1895344 ATR Inhibitor Combined With Stereotactic Body Radiation Therapy and Pembrolizumab for Recurrent Head and Neck Squamous Cell Carcinoma
Brief Title: Testing the Addition of an Anti-cancer Drug, BAY 1895344, With Radiation Therapy to the Usual Pembrolizumab Treatment for Recurrent Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-07522; NCI-2020-07522 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PRO00107885; 10405 (Other: UPMC Hillman Cancer Center LAO); 10405 (Other: CTEP); UM1CA186690 (NIH)
Record Dates: First submitted 2020-10-03; First posted 2020-10-06 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Clinical Stage III HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage IV HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Recurrent Cutaneous Squamous Cell Carcinoma of the Head and Neck; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Paranasal Sinus Squamous Cell Carcinoma; Recurrent Salivary Gland Carcinoma; Stage III Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage III Hypopharyngeal Carcinoma AJCC v8; Stage III Laryngeal Cancer AJCC v8; Stage III Lip and Oral Cavity Cancer AJCC v8; Stage III Major Salivary Gland Cancer AJCC v8; Stage III Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage III Sinonasal Cancer AJCC v8; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck AJCC v8; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Major Salivary Gland Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8; Stage IV Sinonasal Cancer AJCC v8; Unresectable Cutaneous Squamous Cell Carcinoma of the Head and Neck; Unresectable Head and Neck Squamous Cell Carcinoma; Unresectable Hypopharyngeal Squamous Cell Carcinoma; Unresectable Laryngeal Squamous Cell Carcinoma; Unresectable Oral Cavity Squamous Cell Carcinoma; Unresectable Oropharyngeal Squamous Cell Carcinoma; Unresectable Paranasal Sinus Squamous Cell Carcinoma; Unresectable Salivary Gland Squamous Cell Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Specimen Handling; BAY 1895344; pembrolizumab; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, BAY 1895344, SBRT) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Starting on day 7, patients also receive BAY 1895344 PO BID on days 7-9 and 14-16 during cycle 1, and before and after each SBRT treatment during cycle 2 for a total of 9 doses. Beginning cycle 2, patients undergo SBRT starting between days 2 and 8 for 3 fractions with 2-3 days between fractions. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan and/or PET-CT scan and collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Elimusertib; Biological: Pembrolizumab; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT and/or PET-CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Drug: Elimusertib — Given PO
  Other Names: ATR Inhibitor BAY1895344; ATR Kinase Inhibitor BAY1895344; BAY 1895344; BAY-1895344; BAY1895344
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; QL2107; RPH 075; RPH-075; RPH075; SCH 900475; SCH-900475; SCH900475
Procedure: Positron Emission Tomography — Undergo PET-CT scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial evaluates the best dose, possible benefits and/or side effects of combination therapy with elimusertib (BAY 1895344), stereotactic body radiation, and pembrolizumab in treating patients with head and neck squamous cell cancer that has come back (recurrent) and cannot be removed by surgery (unresectable). BAY 1895344 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving BAY 1895344, stereotactic body radiation therapy in combination with pembrolizumab may shrink or stabilize head and neck squamous cell cancer for longer than treatment with radiation and immunotherapy without BAY 1895344.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of BAY 1895344 with concurrent head and neck stereotactic body radiation therapy (SBRT) reirradiation and pembrolizumab.

II. To determine the recommended phase 2 dose (RP2D) of BAY 1895344 in combination with concurrent head and neck SBRT and pembrolizumab.

SECONDARY OBJECTIVE:

I. To observe and record anti-tumor activity (overall response rate, progression-free survival, and overall survival) of BAY 1895344, SBRT, and pembrolizumab for recurrent head and neck squamous cell carcinoma (HNSCC).

EXPLORATORY OBJECTIVE:

I. To identify predictive biomarkers of response to BAY 1895344, SBRT, and pembrolizumab, including, but not limited to the following: genetic alterations of ATM and other deoxyribonucleic acid (DNA) damage response genes, tumor mutational load, circulating tumor DNA, baseline tumor ATM mutation status, tumor PD-L1 expression, and change in circulating Ki67+ CD8+ T-cells relative to baseline.

OUTLINE: This is a dose-escalation study of BAY 1895344 and stereotactic body radiation therapy (SBRT) given with fixed-dose pembrolizumab.

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of each cycle. Starting on day 7, patients also receive BAY 1895344 orally (PO) twice daily (BID) on days 7-9 and 14-16 during cycle 1, and before and after each SBRT treatment during cycle 2 for a total of 9 doses. Beginning cycle 2, patients undergo SBRT starting between days 2 and 8 for 3 fractions with 2-3 days between fractions. Treatment repeats every 21 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scan and/or positron emission tomography (PET)-CT scan and collection of blood samples throughout the trial.

After completion of study treatment, patients are followed up every 13 weeks for at least 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed recurrent or metachronous (second primary), unresectable head and neck squamous cell carcinoma, including oral cavity, oropharynx, larynx, hypopharynx, cutaneous, salivary gland, paranasal sinus, or cervical lymphadenopathy (head and neck cancer of unknown primary). Core needle biopsy (preferably at least three 18-gauge cores) or incisional biopsy is preferred over fine needle aspiration (FNA) for diagnosis of recurrent disease or new primary head and neck squamous cell carcinoma to provide sufficient tumor tissue for correlative studies. Unresectable refers both to patients who have declined surgery and patients deemed unresectable by otolaryngology. This includes patients for whom curative resection is medically contraindicated and/or would be associated with excessive surgical risk (as deemed by the consulting otolaryngologist) or undue surgical morbidity (e.g., total glossectomy, laryngectomy, and/or major resection requiring free flap reconstruction)
* Patients must have either recurrent disease or a new primary squamous cell carcinoma of the head and neck within a previously irradiated area (radiotherapy to dose >= 40 Gy, i.e., in-field recurrence)
* Patients must have completed prior radiotherapy >= 6 months prior to enrollment
* Patients must meet at least one of the following criteria: 1) received prior platinum-containing chemotherapy; and/or 2) tumor expresses PD-L1 (Combined Positive Score [CPS] >= 1)
* Patients who have received anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy must have had disease progression while on this therapy. Patients who have not received prior anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy are also eligible
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of BAY 1895344 with pembrolizumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 50%) and a life expectancy of >= 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >= 9 g/dL or 5.6 mmol/L without transfusion or erythropoietin dependency (within 7 days of assessment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (If total bilirubin > 1.5 x ULN, direct bilirubin must be < ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (=< 5 x ULN for patients with liver metastases)
* Creatinine OR measured or calculated creatinine clearance (CrCl) < 1.5 x institutional ULN OR glomerular filtration rate (GFR) > 60 mL/min/1.73 m^2

  * CrCl should be calculated per institutional standard
* Albumin > 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Patients must have measurable disease (at least one measurable lesion) as per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Baseline imaging must include neck CT (preferably contrast-enhanced) and chest CT or skullbase to midthigh PET/CT (preferably with contrast-enhanced neck CT if diagnostic contrast-enhanced neck CT not available). Patients who have undergone surgery aside from biopsy may be included if gross disease is present within the surgical resection bed or at another site
* Patients must have no contraindications to pembrolizumab, including no history of organ allograft transplantation or active autoimmune disease (active defined as having autoimmune disease-related symptoms and detectable autoantibodies) that has required systemic treatment in the past 2 years (i.e., use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Human immunodeficiency virus (HIV)-infected patients may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * They must have a CD4 count of greater than 250 cells/mcL
  * They must not be receiving prophylactic therapy for an opportunistic infection
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy (e.g., not hepatitis B surface antigen [HBsAg] reactive), if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load (e.g., HCV ribonucleic acid [RNA] [qualitative] is not detected)
* Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging using the identical imaging modality for each assessment, either magnetic resonance imaging [MRI] or computed tomography [CT] scan, for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial (e.g. basal cell carcinoma, early-stage differentiated thyroid carcinoma, low-risk prostate cancer, ductal carcinoma in situ of the breast, squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer). Patients with 10 or fewer distant metastases may be eligible for this trial if they meet performance status inclusion criteria
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better
* Enrolling site must perform PD-L1 testing on tumor biopsy per institutional protocol (local testing or tissue sent to outside laboratory for PD-L1 immunohistochemistry (IHC) 22C3 pharmDx). Combined positive score (CPS) is recommended for PD-L1 scoring. Test result does not need to be available at the time of enrollment and treatment initiation, unless the patient has not received prior platinum-containing chemotherapy. For patients without a history of platinum-containing chemotherapy, PD-L1 testing with CPS >= 1 is required to be eligible to receive pembrolizumab
* Female patients of childbearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. The effects of BAY 1895344 on the developing human fetus are unknown. For this reason and because DNA-damage response inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months after completion of BAY 1895344 therapy or 4 months after completion of pembrolizumab therapy, whichever is later. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of BAY 1895344 therapy or 4 months after completion of pembrolizumab therapy, whichever is later

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible

Exclusion Criteria:

* Patients who are unable to take oral medications
* Patients with nasopharyngeal carcinoma, paranasal sinus cancers with histology other than squamous cell carcinoma, or salivary gland cancers with histology other than squamous cell carcinoma
* Patients who have had more than one prior course of head and neck radiotherapy
* Patients who have disease surrounding >= 180 degrees of the carotid artery
* Patients with gross tumor involvement of the mandible
* Patients with widely metastatic disease.

  * Note: Patients with oligometastatic disease (defined as ten or fewer distant metastases) may qualify for the study
* Patients who have had chemotherapy, targeted small-molecule therapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study

  * Note: Patients with =< grade 2 neuropathy or =< grade 2 alopecia are an exception to this criterion and may qualify for the study
  * Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients who are currently participating and receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including granulocyte colony-stimulating factor [G-CSF], granulocyte macrophage colony-stimulating factor [GM-CSF], or recombinant erythropoietin) within 4 weeks prior to initiating the study drug BAY 1895344
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the study principal investigator (PI)
* Has had a prior monoclonal antibody other than anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events (AEs) due to agents administered more than 4 weeks earlier.

Note: Patients who received anti-PD-1, anti-PD-L1, or anti-PD-L2 therapy within 4 weeks prior to study initiation are eligible if they have exhibited disease expression while on this therapy

* Has new or progressive brain metastases, or leptomeningeal disease
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, in situ cervical cancer, ductal carcinoma in situ of the breast, early-stage differentiated thyroid cancer, or low-risk prostate cancer. Note: As discussed above, patients with limited metastatic disease (10 or fewer distant metastases) may qualify for the study
* Patients with carcinomatous meningitis should be excluded
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 1893544 or pembrolizumab
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Patients whose disease has improved or remained stable (no evidence of disease progression) while receiving therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent are ineligible
* Patients receiving any medications that are substrates of CYP3A4 with a narrow therapeutic window, or strong inhibitors/inducers of CYP3A4 are ineligible, if they cannot be transferred to alternative medication. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because BAY 1895344 as a DNA-damage response inhibitor may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 1895344, breastfeeding should be discontinued if the mother is treated with BAY 1895344 and for 4 months after the end of BAY 1895344 treatment. These potential risks may also apply to other agents used in this study
* Has a known history of active tuberculosis (TB)
* Has received a live vaccine within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted. Similarly, coronavirus disease 2019 (COVID-19) vaccines are permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2024-11-27 (Actual); Study Completion 2025-12-11 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose of elimusertib (BAY 1895344) and concurrent stereotactic body radiation therapy (Dose Escalation Phase) | Within 90 days of treatment initiation
Incidence of late adverse events (Dose Expansion Phase) | Within 1 year of treatment initiation
  Will be assessed per Common Terminology Criteria for Adverse Events (CTCAE) version 5.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 12 months
  Will be assessed per CTCAE version 5. The frequency and percentage of adverse events will be provided overall and by dose level for any grade and attribution as well as for grade 3 or greater adverse events, at least possibly related to treatment.
Locoregional control | Up to 2 years
  A competing risk analysis will be conducted with local failure, distal failure, and death as competing events. The cumulative incidence and 95% confidence interval for local failure will be estimated. Time to each event will be measured from the start of treatment regimen (day 1 pembrolizumab).
Progression-free survival | From the start of treatment regimen (day 1 pembrolizumab) until documented local or distal failure or death from any cause, assessed up to 2 years
  Will be estimated using the method of Kaplan-Meier.
Overall response rate | Up to 2 years
  Defined as a complete response or partial response based on the Response Evaluation Criteria in Solid Tumors 1.1 criteria. The proportion of patients responding to the treatment regimen and corresponding 95% confidence interval estimates will be calculated.
1-year overall survival | From the start of treatment regimen (day 1 pembrolizumab) until death from any cause, assessed up to 1 year
  Will be estimated using the method of Kaplan-Meier.
Quality of life | At 3, 6, and 12 months from start of treatment
  Will be assessed by the Functional Assessment of Cancer Therapy for Patients With Head and Neck Cancer, version 4. The frequency and percentage of responses to the quality of life questionnaire will be summarized at 3, 6, and 12 months post-treatment and interpreted descriptively.

OTHER OUTCOMES:
Potential predictive biomarkers of response | Up to 2 years
  Will investigate the association between potential predictive biomarkers of response to treatment. Tumor mutation burden will be categorized as high (above median) or low (equal to or below median). Other biomarker expression levels will be categorized as high versus absent/reduced. The chi-square or Fisher exact test will be used to study associations between expression levels and tumor response (complete response/partial response; stable/progressive disease). Associations with time-to-event endpoints will be investigated using the log rank test. Differences in change in circulating Ki67+ CD8+ T-cells relative to baseline between levels of tumor response will be explored using the t-test or non-parametric equivalent (e.g., Mann-Whitney) if appropriate. Cox regression will be used to explore associations between change in in circulating Ki67+ CD8+ T-cells and time-to-event endpoints. Other biomarkers will be analyzed similarly.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne M Mowery, Principal Investigator — University of Pittsburgh Cancer Institute LAO
Locations (11):
- United States (11):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm